CLINICAL TRIAL: NCT03505983
Title: Criteria for Advanced Prosthetic Foot Prescription
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); James A. Haley Veterans Administration Hospital (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Maikos, Director, VISN 2 Gait and Motion Analysis Laboratory, VA New York Harbor Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB #01603; CDMRP-OP150095 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2018-03-07; First posted 2018-04-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Prosthesis User; Amputation; Traumatic, Limb, Lower
Keywords: Prosthetic Limb Design; Prosthesis Fitting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor and statistician will be blinded to foot type during data processing and analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Articulating ESR Prosthetic Foot First (Active Comparator): Subjects will start with an Articulating ESR prosthetic foot first for 1 week, then will complete an additional week with the ESR prosthetic foot, and a powered prosthetic foot for 1 week.The final 4 weeks, all prosthetic feet will be available for use and subjects will self-select which foot to use for daily activities.
  Interventions: Device: Articulating ESR Prosthetic Foot First
- Powered Prosthetic Foot First (Active Comparator): Subjects will start with a powered prosthetic foot first for 1 week, then will complete an additional week with an articulating ESR prosthetic foot and an ESR prosthetic foot for 1 week. The final 4 weeks, all prosthetic feet will be available for use and subjects will self-select which foot to use for daily activities.
  Interventions: Device: Powered Prosthetic Foot First
- ESR Prosthetic Foot First (Active Comparator): Subject will start with an energy storing and returning (ESR) prosthetic foot first for 1 week, then will complete an additional week with an articulating ESR prosthetic foot, and a powered prosthetic foot for 1 week. During the final 4 weeks of the study, all prosthetic feet will be available and subjects can self-select which foot to use.
  Interventions: Device: ESR Prosthetic Foot First

INTERVENTIONS:
Device: ESR Prosthetic Foot First — Subjects will start with an ESR foot first for 1 week, then will complete an additional week with an articulating ESR foot and a powered foot for 1 week. The final 4 weeks of the study, all prosthetic feet will be available and subjects can self-select which foot to use.
  Arms: ESR Prosthetic Foot First
Device: Articulating ESR Prosthetic Foot First — Subjects will start with an articulating ESR foot first for 1 week, then will complete an additional week with an articulating ESR foot and a powered foot for 1 week. The final 4 weeks of the study, all prosthetic feet will be available and subjects can self-select which foot to use.
  Other Names: Odyssey (College Park); Elan (Endolite); MotionFoot (Fillauer); Proflex (Ossur); Echelon (Endolite); Tribute (College Park); Proprio (Ossur); TruStep (College Park); Kinterra (Freedom Innovations); Flex Foot Balance with DP Flexion (Ossur); Raize (Fillauer); Echelon VT (Endolite); Triton Smart Ankle (Otto Bock); Venture (College Park); Kinnex (Freedom Innovations)
  Arms: Articulating ESR Prosthetic Foot First
Device: Powered Prosthetic Foot First — Subjects will start with a powered prosthetic foot first for 1 week, then will complete an additional week with an articulating ESR foot and an ESR foot for 1 week. The final 4 weeks of the study, all prosthetic feet will be available and subjects can self-select which foot to use.
  Other Names: emPOWER (Otto Bock)
  Arms: Powered Prosthetic Foot First

SUMMARY:
The purpose of this study is to develop criteria for prosthetic foot prescription for Veterans and Service Members with transtibial limb loss. The objectives are to: 1) Determine the appropriate functional outcome tests and measures to support the prescription of a type of Energy Storing and Returning (ESR) non-articulating, articulating or active plantarflexion prosthetic ankle-foot for a Veteran or Service Member with transtibial limb loss. 2) Correlate patient goals and subjective measures with objective data to determine the appropriate prosthetic ankle-foot category that will facilitate the greatest overall function to the user. 3) Develop criteria for the appropriate prescription of non-articulating ESR, articulating ESR, and active plantar flexion ESR ankle-foot units.

ELIGIBILITY:
Inclusion Criteria:

* DEERS eligible Veteran or Service Member, or civilian with unilateral transtibial amputation
* Currently using an Energy Storing and Returning prosthetic foot with a well-fitting socket as a primary or back-up prosthesis
* Achieved a "Modified Independence" score on the Functional Independence Measure (FIM) for the locomotion mobility items
* Has a minimum clearance of 8 ¾ inches to accommodate all feet

Exclusion Criteria:

* Has active wounds/ulcers or significant musculoskeletal comorbidities on their intact limb that would impair their ability to participate in all functional outcome measures
* Has any comorbidity that results in rapid limb volume changes (i.e. end stage renal disease with dialysis),
* Weighs more than 275 pounds, the maximum product weight load
* Is unable or unwilling to comply with all research visits
* Has cognitive deficit(s) or mental health pathology limiting a subject's ability to participate fully in the study
* Women who are pregnant or plan to become pregnant during study activities. This will be determined by asking the participant if they are pregnant or if they believe that they may be pregnant. This question will only be asked at inclusion, as biomechanical changes will only be impacted if the woman is in the 2nd or 3rd trimester, and will not be impacted if the participant becomes pregnant while in the study.
* Poorly fitting socket
* Vision loss that requires use of an assistive device for gait
* Upper Limb Amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 6-min walk distance for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The 6-minute walk test measures the distance an individual can walk in 6 minutes without help or encouragement.
Change in TUG times for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The TUG measures the time taken by an individual to stand up from a standard arm chair, walk a distance of 10 feet, turn, walk back to the chair, and sit down.
Change in 4SST times for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The four-square step test is a higher order complex task assessing dynamic balance.
Change in AmpPRO for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The AmpPro is a 21-item instrument designed to measure basic prosthetic mobility of individuals with lower extremity amputation.
Change in Stair Assessment Index (SAI) for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The SAI is a rated qualitative scale on how an individual with lower limb amputation negotiates up and down a staircase.
Change in Hill Assessment Index (HAI) for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The HAI is a rated qualitative scale on how an individual with lower limb amputation negotiates up and down a ramp.
Change in Gait Evaluation for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  Biomechanical evaluation of gait.

SECONDARY OUTCOMES:
Change in Prosthetic Evaluation Questionnaire (PEQ) score for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The PEQ is a self-report Visual Analog Scale questionnaires for persons with lower limb amputations who use a prosthesis. It consists of 9 validated subscales. They are used to evaluate the prosthesis and life with the prosthesis. Most questions in the PEQ use a visual analog scale format. Each visual analog scale is scored as a continuous numerical variable measured as the distance in millimeters from the left endpoint of the line to the point at which the respondent's mark crosses the line. Each line is 100 mm long and is always measured from the left (0-100). The questions are all worded so that a higher number (toward the right) will correspond with a more positive response. Subscale scores are calculated by computing the average (arithmetic mean) of all the questions which make up that particular scale. Only subscales are calculated. A total combined score is not calculated.
Change in Short Form (SF)-12 for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The SF-12 is a questionnaire used to measure the relationship between physical and mental health functioning and the social determinants of health. It is a self-reported questionnaire, on a rating scale, called a Likert Scale. The participant taking this questionnaire will check one response box per question. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Age-specific mean difference score (difference score) is calculated and is the amount by which a person's score differs from their age group's mean score. By looking at difference scores, it is clear whether a person is more or less healthy than other persons in his or her comparison group.
Change in OPUS for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  OPUS is a set of self-report instruments that assess functional status, quality of life, and satisfaction with devices and services that can be used in an orthotics and prosthetics clinic. The OPUS Health Quality of Life Score is the sum of the scores for the 23 items (0 - 92). The OPUS lower extremity total score is the sum of the scores for the 20 items (0 - 80). OPUS Satisfaction With Device Score is the sum of the scores for items 1-11 (11 - 55). Satisfaction With Services Score is the sum of the scores for items 12-21 (10 - 50). A higher score indicates a better outcome for all measures.
Final Visit Guided Interview | Administered one time at Final Visit, which will occur 7 weeks after enrollment.
  Final Visit questionnaire to evaluate subjective preferences. This is a free response questionnaire, in which the participant can answer in open-ended format.
Change in responses to Prosthetic Evaluation Questionnaire-Addendum (PEQ-A) for each prosthetic foot type | Once per week, at Week 1, Week 2, and Week 3 after enrollment
  The PEQ-A is a free response 2-question questionnaire, in which the participant is asked whether and how many times they had experienced a fall or near-fall in the previous week using the particular prosthetic foot.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Maikos, PhD, Principal Investigator — Director, VISN 2 Gait and Motion Analysis Laboratory
Locations (1):
- VA New York Harbor Healthcare System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maikos JT, Hendershot BD, Pruziner AL, Hyre MJ, Chomack JM, Phillips SL, Heckman JT, Sidiropoulos AN, Dearth CL, Nelson LM. Criteria for Advanced Prosthetic Foot Prescription: Rationale, Design, and Protocol for a Multisite, Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 4;12:e45612. doi: 10.2196/45612. PMID 37014672